CLINICAL TRIAL: NCT00041652
Title: A Phase I/II Clinical Trial of Immunotherapy With Humanized MN-14 IgG in Recurrent, Metastatic, Unresectable Colorectal and Breast Carcinomas
Brief Title: Safety Study of hMN14 to Treat Either Colorectal or Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hMN14-04
Record Dates: First submitted 2002-07-11; First posted 2002-07-15 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2005-10

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Breast Cancer; Breast Neoplasms
Keywords: Colorectal Cancer; Colon Cancer; Rectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Breast Neoplasms | interventions — labetuzumab

INTERVENTIONS:
Drug: hMN14 (labetuzumab)

SUMMARY:
The purpose of this trial is to determine the safety of hMN14 at different dose levels in the treatment of either colorectal or breast cancer.

ELIGIBILITY:
Disease Characteristics:

* Histologic or cytologic diagnosis or either, colonic, rectal, or breast carcinoma
* Measurable lesion diagnosed by CT scan
* Recurrent/metastatic disease considered surgically unresectable.

Prior/Concurrent Therapy:

* Chemotherapy: Patients who either have failed at least one regimen of standard systemic therapy, or are clinically asymptomatic and are not presently being considered for chemotherapy (Enrollment must occur at least 4 weeks beyond last treatment)
* Other: Prior treatment with investigational agents is excluded unless follow-up is completed and patient is off study

Patient Characteristics/Inclusion Criteria:

* Performance Status: Patients with a Karnofsky performance status > 70% (or equivalent, ECOG 0-1) and expected survival of at least 3 months.
* Hematopoietic: WBC >/= 3000 mm3, neutrophils >/= 1500 mm3, platelets >/= 75,000, CEA < 300 ng/mL
* Hepatic: Serum bilirubin </= 2.0 mg/dL, ALT < 2.5 x IULN
* Cardiovascular: Patients with LVEF >/= 40% by required MUGA/2D-ECHO study.
* Pulmonary: Patients with FEV1 >/= 60% by required Pulmonary Function Tests
* Other: Patients agreeing to use a medically effective method of contraception during and for a period of 3 months after the treatment period. A pregnancy test will be preformed on each premenopausal female of childbearing potential immediately prior to entry into the study. Patients able to understand and give written informed consent. Patients with a significant concurrent medical condition that could affect the patient's ability to tolerate or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2000-02; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Terence Rugg, MD, Study Director — Gilead Sciences; Lauri Welles, MD, Study Chair — Gilead Sciences
Locations (1):
- Hoag Cancer Center, Newport Beach, California, United States